CLINICAL TRIAL: NCT00779259
Title: A Pharmacokinetic Drug-Drug Interaction Study to Evaluate the Effect of Steady-State Quinine Sulfate on the Pharmacokinetics of Single-Dose Theophylline in Healthy Adult Males
Brief Title: Drug - Drug Interaction Study Between Quinine Sulfate and Theophylline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-001-07-1002; R07-0738
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
Keywords: quinine sulfate; theophylline; drug interactions; cytochrome p450; humans; male; adult
MeSH Terms: interventions — Theophylline; Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Theophylline alone (Active Comparator): baseline theophylline pharmacokinetics
  Interventions: Drug: Theophylline 300mg
- Quinine alone (Active Comparator): baseline quinine pharmacokinetics at steady state
  Interventions: Drug: Quinine 648 mg
- Theophylline with steady state quinine (Experimental): Theophylline pharmacokinetics in the presence of steady state quinine and quinine pharmacokinetics in the presence of theophylline.
  Interventions: Drug: Theophylline 300 mg; Drug: Quinine 648 mg

INTERVENTIONS:
Drug: Theophylline 300mg — Single doses of theophylline 300 mg as an immediate-release oral solution 80mg/15ml concentration administered alone at 7 am on Day 1 after an overnight fast of at least 10 hours and along with quinine sulfate (2 x 324 mg capsules) at 7am on Day 12 after an overnight fast of at least 10 hours.
  Arms: Theophylline alone
Drug: Quinine 648 mg — 648 mg quinine sulfate(2 x 324 mg capsules) initiated at 3pm on Day 5 and taken every 8 hours through Day 11 and co-administered with theophylline 300 mg as an immediate-release oral solution 80 mg/15 ml concentration at 7am on Day 12.
  Arms: Quinine alone
Drug: Theophylline 300 mg — Single doses of theophylline 300 mg as an immediate-release oral solution 80mg/15ml concentration administered alone at 7 am on Day 1 after an overnight fast of at least 10 hours and along with quinine sulfate (2 x 324 mg capsules) at 7am on Day 12 after an overnight fast of at least 10 hours.
  Arms: Theophylline with steady state quinine
Drug: Quinine 648 mg — 648 mg quinine sulfate(2 x 324 mg capsules) initiated at 3pm on Day 5 and taken every 8 hours through Day 11 and co-administered with theophylline 300 mg as an immediate-release oral solution 80 mg/15 ml concentration at 7am on Day 12.
  Arms: Theophylline with steady state quinine

SUMMARY:
In a prior in vitro study using human hepatocytes quinine was shown to induce the activity of Cytochrome p450 CYP 1A2. The present study will evaluate the extent to which quinine sulfate-related induction of this enzyme effects the pharmacokinetics of theophylline, a sensitive probe drug for the activity of CYP 1A2. It will also evaluate the effect of single-dose theophylline on the pharmacokinetics of steady-state quinine sulfate.

DETAILED DESCRIPTION:
This study will evaluate the effect of steady-state quinine sulfate on the pharmacokinetics of single dose theophylline and the effect of single dose theophylline on the pharmacokinetics of steady-state quinine sulfate in healthy adult males under fasting conditions. In this non-blinded, crossover study 24 normal, healthy, non-smoking, non-obese male volunteers will serve as their own controls in two cohorts, one consisting of 8 subjects and one consisting of 16 subjects. On Day 1 after a minimum overnight fast of 10 hours, the 8 study participants in cohort 1 will receive a single oral dose of theophylline (300 mg as an immediate-release oral solution 80 mg/ 15 ml concentration). After a 4 day washout period, the 8 subjects will receive a 648 mg dose of quinine sulfate (2 x 324 mg capsules) every 8 hours (dosing at 7 am, 3 pm and 11 pm daily) beginning with the 3 pm dose on Day 5 and continuing through the morning dose on Day 12. The 8 subjects will be co-administered single oral doses of theophylline (300 mg as an immediate-release oral solution 80 mg/ 15 ml concentration) and quinine sulfate (2 x 324 mg capsules) at 7 am on Day 12. Cohort 2 will be dosed on the basis of safety findings in Cohort 1. If ≥ 50% of the volunteers in cohort 1 do not tolerate the 648 mg dose of quinine sulfate, the second cohort of 16 volunteers will receive a dose of quinine sulfate reduced from 648 mg to 324 mg every 8 hours. In each cohort serial pharmacokinetic blood samples will be drawn at times sufficient to adequately define the pharmacokinetics of theophylline and quinine. Blood samples for the measurement of theophylline plasma concentrations will be collected on Days 1 and 12 prior to dosing and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose. Blood samples for the measurement of quinine sulfate plasma concentrations will be collected on Day 11 prior to the morning dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, and 8 hours post dose and on Day 12 prior to dosing and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6 and 8 hours post-dose. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vital signs (sitting blood pressure and pulse) will be measured prior to the morning dose and at 1, 2 and 4 hours after administration of the morning dose on Days 1, 11 and 12. On Day 5, sitting blood pressure and pulse will be measured prior to the afternoon dose and at 1, 2 and 4 hours after administration of the afternoon dose. ECGs will be collected pre-dose and at 4 hours after the morning dose on study Days 1, 5, 11 and 12. All adverse events whether elicited by query, spontaneously reported or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy non-smoking, non-obese (≥ 55kg and within 15% of ideal body weight) adult male volunteers 18-45 years of age

Exclusion Criteria:

* Subjects with history or presence of glucose 6 phosphate dehydrogenase deficiency, myasthenia gravis, optic neuritis, glaucoma or significant cardiovascular disease (including hypotension, bradycardia or EKG abnormalities), pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease or an active sexually transmitted disease
* Subjects with significant blood loss in the prior 56 days, plasma donation within 7 days , hemoglobin <12.0 g/dl or who have participated in another clinical trial within the prior 30 days
* Subjects with recent (2-year) history or evidence of alcoholism or drug abuse
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome P450 (CYP) enzymes and/or P-glycoprotein within 30 days prior to the first dose and throughout the study
* Subjects who test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV).
* Subjects who are pregnant or lactating or have hypersensitivity to quinine sulfate, mefloquine, quinidine or hypersensitivity to theophylline or aminophylline.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Study Chair — Mutual Pharmaceutical; Barrie March, MD, Principal Investigator — PRACS Institute
Locations (1):
- PRACS Institute, Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking, adult male volunteers from the community at large were enrolled.
Pre-assignment Details: Fifty-two (52) subjects were screened. Ten (10) were screen failures, eight (8) did not return and ten (10) were discharged.
Groups:
- Theophylline Alone, Quinine Alone, Theophylline With Quinine: This study was done in two cohorts, each receiving the same dosing regimen. For each cohort, all subjects received a single dose of theophylline (300 mg as an immediate-release oral solution 80 mg/15 ml concentration) at 7:00am on Day 1 following an overnight fast of at least 10 hours. After a 4-day washout period, subjects received 648 mg of quinine sulfate (2 x 324 mg capsules) every 8 hours (dosing occurred at 7am, 3pm and 11pm daily) starting with the 3pm dose on Day 5 and continuing through the morning dose on Day 12. Subjects also received a single 300 mg dose of theophylline along with their 648 mg quinine sulfate dose on the morning of Day 12.
Period: Theophylline Alone
Arm/Group | Theophylline Alone, Quinine Alone, Theophylline With Quinine
Started | 24
Completed | 24
Not Completed | 0
Period: 4 Day Washout Period
Arm/Group | Theophylline Alone, Quinine Alone, Theophylline With Quinine
Started | 24
Completed | 24
Not Completed | 0
Period: Quinine Alone
Arm/Group | Theophylline Alone, Quinine Alone, Theophylline With Quinine
Started | 24
Completed | 22
Not Completed | 2
Not completed — Adverse Event | 2
Period: Theophylline With Quinine
Arm/Group | Theophylline Alone, Quinine Alone, Theophylline With Quinine
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Theophylline Alone, Quinine Alone, Theophylline With Quinine
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 23
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.25 (6.038)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration(Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: Serial pharmacokinetic blood samples for theophylline collected on Days 1 and 12 before dosing and for 48 hours post-dose. Serial pharmacokinetic blood samples for quinine collected on Days 11 and 12 before dosing and for 8 hours after the morning dose.
Population: A total of 24 healthy adult male subjects participated in this study, 22 of whom completed. Pharmacokinetic analyses of theophylline are based on 19 subjects (data for 2 subjects excluded due to vomiting post-dose and for 1 subject as an outlier. Pharmacokinetic analyses of quinine are based on 20 subjects (excluding the two who vomited).
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Theophylline Alone: At 7am on Day 1 after a fast of at least 10 hours, all subjects received a single dose of theophylline (300 mg as an immediate-release oral solution 80mg/15ml concentration)followed by a 4-day washout period.
- Quinine Alone: On Day 5 in the afternoon, dosing of quinine sulfate (2 x 324 mg capsules) was initiated and continued every 8 hours without regard to meals through Day 11.
- Theophylline in the Presence of Quinine; Quinine in the Presence of Theophylline: At 7am on Day 12 after a fast of at least 10 hours, subjects received a single dose of theophylline (300 mg as an immediate-release oral solution 80mg/15ml concentration) and quinine sulfate (2 x 324 mg capsules).
Arm/Group | Theophylline Alone | Quinine Alone | Theophylline in the Presence of Quinine | Quinine in the Presence of Theophylline
Number analyzed (Participants) | 19 | 20 | 19 | 20
ug/mL | 9.58 (1.66) | 6.63 (1.63) | 9.81 (1.35) | 7.47 (1.77)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve beginning from the first dose (time 0) to the last measurable concentration (time t), as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug-hr/mL
Groups:
- Theophylline Alone: At 7am on Day 1 after a fast of at least 10 hours, all subjects received a single dose of theophylline (300 mg as an immediate-release oral solution 80mg/15ml)followed by a 4 day washout period
- Theophylline in Presence of Quinine; Quinine in Presence of Theophylline: At 7am on Day 12 after a fast of at least 10 hours, subjects received a single dose of theophylline (300 mg as an immediate-release oral solution 80mg/15ml) and quinine sulfate (2 x 324 mg capsules).
Arm/Group | Theophylline Alone | Quinine Alone | Theophylline in Presence of Quinine | Quinine in Presence of Theophylline
Number analyzed (Participants) | 19 | 20 | 19 | 20
ug-hr/mL | 103.47 (35.82) | 45.17 (11.41) | 92.72 (31.17) | 51.68 (13.11)

3. Primary Outcome: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)].
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞)was calculated as the sum of the AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: Serial pharmacokinetic blood samples for theophylline collected on Days 1 and 12 before dosing and for 48 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug-hr/mL
Arm/Group | Theophylline Alone | Theophylline in Presence of Quinine
Number analyzed (Participants) | 19 | 19
ug-hr/mL | 108.21 (37.33) | 96.88 (31.95)

4. Secondary Outcome: Electrocardiogram (ECG) Evaluation of the Maximum QT Interval Corrected for Heartrate (QTc), Quinine Study Day 11.
Description: The QT interval assesses cardiac repolarization and risk for arrhythmias. It is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. QTc is the QT interval corrected for heartrate.
Time Frame: 5 hours - measured 1 hour pre-dose and then at 4 hours after the morning dose on Day 11
Measure: Number; unit: msec
Groups:
- 1 Hour Before Morning Dose of Quinine on Study Day 11: measured 1 hour prior to the morning dose of Quinine on study Day 11
- 4 Hours After Morning Dose of Quinine on Study Day 11: measured 4 hours after the morning dose of quinine
Arm/Group | 1 Hour Before Morning Dose of Quinine on Study Day 11 | 4 Hours After Morning Dose of Quinine on Study Day 11
Number analyzed (Participants) | 23 | 23
msec | 453.33 | 451.33

5. Secondary Outcome: Electrocardiogram (ECG) Evaluation of the Maximum QT Interval Corrected for Heartrate (QTc), Theophylline Co-administered With Quinine, Study Day 12.
Description: as for outcome 4
Time Frame: 5 hours - measured 1 hour pre-dose and then at 4 hours post-dose on Day 12
Measure: Number; unit: msec
Groups:
- 1 Hour Before Co-Administered Dose of Theophylline/Quinine: measured 1 hour prior to the 7 am co-administered dose of theophylline and quinine
- 4 Hours After Co-Administered Dose of Theophylline/Quinine: measured 4 hours after the 7 am co-administered dose of theophylline and quinine
Arm/Group | 1 Hour Before Co-Administered Dose of Theophylline/Quinine | 4 Hours After Co-Administered Dose of Theophylline/Quinine
Number analyzed (Participants) | 22 | 22
msec | 452 | 455.33

ADVERSE EVENTS:
Groups:
- Theophylline Alone: At 7am on Day 1 after a fast of at least 10 hours, all subjects received a single dose of theophylline (300 mg as an immediate-release oral solution 80 mg/15 ml)followed by a 4 day washout period
- Theophylline Co-administered With Quinine: At 7am on Day 12 after a fast of at least 10 hours, subjects received a single dose of theophylline (300 mg as an immediate-release oral solution 80 mg/15 ml) and quinine sulfate (2 x 324 mg capsules).
Arm/Group | Theophylline Alone | Quinine Alone | Theophylline Co-administered With Quinine
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 0
Other Adverse Events (participants affected / at risk) | 7 | 22 | 20
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Theophylline Alone | Quinine Alone | Theophylline Co-administered With Quinine
drug hypersensitivity (General disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Theophylline Alone | Quinine Alone | Theophylline Co-administered With Quinine
palpitations (Cardiac disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
deafness (Ear and labyrinth disorders) | 0/24 (0) | 2/24 (2) | 1/24 (1)
deafness bilateral (Ear and labyrinth disorders) | 0/24 (0) | 2/24 (2) | 0/24 (0)
dysacusis (Ear and labyrinth disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
ear discomfort (Ear and labyrinth disorders) | 0/24 (0) | 7/24 (7) | 0/24 (0)
ear pain (Ear and labyrinth disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
hearing impaired (Ear and labyrinth disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
hypoacusis (Ear and labyrinth disorders) | 0/24 (0) | 3/24 (3) | 0/24 (0)
tinnitus (Ear and labyrinth disorders) | 0/24 (0) | 13/24 (13) | 0/24 (0)
abdominal pain upper (Gastrointestinal disorders) | 0/24 (0) | 1/24 (1) | 1/24 (1)
diarrhea (Gastrointestinal disorders) | 1/24 (1) | 1/24 (1) | 0/24 (0)
haematochezia (Gastrointestinal disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
nausea (Gastrointestinal disorders) | 1/24 (1) | 5/24 (5) | 12/24 (12)
retching (Gastrointestinal disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
stomach discomfort (Gastrointestinal disorders) | 0/24 (0) | 2/24 (2) | 0/24 (0)
vomiting (Gastrointestinal disorders) | 0/24 (0) | 0/24 (0) | 2/24 (2)
chest discomfort (Gastrointestinal disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
chest pain (General disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
chills (General disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
feeling cold (General disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
feeling hot (General disorders) | 0/24 (0) | 2/24 (2) | 2/24 (2)
feeling jittery (General disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
pallor (General disorders) | 0/24 (0) | 1/24 (1) | 3/24 (3)
pyrexia (General disorders) | 0/24 (0) | 2/24 (2) | 0/24 (0)
heart rate increased (Investigations) | 0/24 (0) | 1/24 (1) | 1/24 (1)
anorexia (Metabolism and nutrition disorders) | 0/24 (0) | 1/24 (1) | 1/24 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0/24 (0) | 0/24 (0) | 2/24 (2)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/24 (0) | 1/24 (1) | 1/24 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
dizziness (Nervous system disorders) | 2/24 (2) | 6/24 (6) | 9/24 (9)
dysgeusia (Nervous system disorders) | 0/24 (0) | 3/24 (3) | 0/24 (0)
headache (Nervous system disorders) | 1/24 (1) | 2/24 (2) | 9/24 (9)
paraesthesia (Nervous system disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
syncope (Nervous system disorders) | 1/24 (1) | 0/24 (0) | 3/24 (3)
tremor (Nervous system disorders) | 0/24 (0) | 0/24 (0) | 2/24 (2)
confusional state (Psychiatric disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
depressed mood (Psychiatric disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
disorientation (Psychiatric disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
restlessness (Psychiatric disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
thinking abnormal (Psychiatric disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
urinary hesitation (Renal and urinary disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 2/24 (2) | 0/24 (0)
drug eruption (Skin and subcutaneous tissue disorders) | 0/24 (0) | 0/24 (0) | 2/24 (2)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
rash (Skin and subcutaneous tissue disorders) | 0/24 (0) | 0/24 (0) | 1/24 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days